CLINICAL TRIAL: NCT05944783
Title: Bioequivalence Studies of Dasatinib 100 Mg Tablets in Healthy Colombian Subjects in Postprandial Condition
Brief Title: Bioequivalence Studies of Dasatinib 100 Mg
Acronym: BE-Dasatinib
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de Atencion e Investigacion Medica (Network)
Responsible Party: Principal Investigator, Humberto Reynales MD MSc PhD, Dr MD MSc PhD, Centro de Atencion e Investigacion Medica
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DASAT-BIO-001-2022; DASAT-BIO-001-2022 (Other: CAIMED)
Record Dates: First submitted 2022-08-11; First posted 2023-07-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Myeloma Multiple
Keywords: Dasatinib , fed condition, bioequivalence
MeSH Terms: conditions — Multiple Myeloma | interventions — Dasatinib

STUDY DESIGN:
Intervention Model Description: Dasatinib bioequivalence study in fed condition
Who Masked: Investigator, Outcomes Assessor
Masking Description: randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liteda® (Active Comparator): Dasatinib 100 mg tablets Lab. Tecnofarma Colombia S.A.S. Liteda®
  Interventions: Drug: Dasatinib 100 MG
- Sprycel® (Active Comparator): Dasatinib 100 mg tablets Lab. Bristol-Myer Squibb Sprycel®
  Interventions: Drug: Dasatinib 100 MG

INTERVENTIONS:
Drug: Dasatinib 100 MG — single dose of 100 mg Dasatinib tablets
  Other Names: sprycel

SUMMARY:
A bioequivalence study of Dasatinib will be carried out in 46 healthy subjects, in fed condition, following the complete replicated design, randomized, comparative of 2 sequences, 2 study formulations, in a single dose of 100 mg of Dasatinib tablets / coated tablets, 4 periods. , with a washout time of 7 days between each dose

DETAILED DESCRIPTION:
A bioequivalence study of Dasatinib in 46 healthy subjects, in fed condition, complete replicated design, comparative of 2 sequences, 2 formulations, single dose of 100 mg of Dasatinib tablets / coated tablets, 4 periods. , with a washout time of 7 days between each dose

ELIGIBILITY:
Inclusion Criteria:

* Men of legal age between 18 to 50 years.
* Have been clinically diagnosed as healthy by the trial doctor.
* Subjects with clinical laboratory results within normal ranges and/or suitable by medical selection.
* Non-smoking subjects for the last 3 months.
* Have signed the informed consent.
* Body mass index between 18-30 kg/m2
* Subject with complete contact information (cell phone and/or contact landline, address, email).
* Subject who has a family member or guardian with a contact telephone number.
* Subject to the availability of time to comply with scheduled visits and activities.

Exclusion Criteria:

* Subject with a diagnosis of renal, cardiac, hepatic, immunological, dermatological, endocrine, gastrointestinal, neurological or psychiatric disease.
* Subjects diagnosed with positive COVID 19
* Subject diagnosed with hematological disorders, such as anemia and/or polycythemia.
* Subjects with a history of gastric surgeries.
* Permanent or temporary use during the last 15 days of any type of medication, both on their own initiative and by medical prescription. Except female patients who are planning regularly with the same contraceptive method in the last 6 months prior to the start of this trial.
* Smoker in the last 3 months, regardless of the number of cigarettes.
* Consumption of xanthines from coffee, tea or chocolate during the previous 48 hours
* Drinker of alcohol in more than 16 grams every week equivalent to 1 beer or 2 glasses of wine during the last 15 days.
* Consumption of drugs of abuse or psychoactive substances reported as a positive test.
* Known hypersensitivity to the active substance or to the excipients of the test product.
* Medical history of angioedema or anaphylaxis.
* Subject diagnosed with human immunodeficiency virus infection, hepatitis B or positive hepatitis C.
* Have participated in clinical studies in the 4 months prior to the start of this trial.
* Have donated blood in the 30 days prior to the start of the trial.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Cmax - Maximum Observed Concentration | 2 days
  Bioequivalence based on Cmax
AUC0-24 - Area Under the Concentration-time Curve From Time Zero to 24 Hours Post-dose | 2 days
  Bioequivalence based on AUC0-24

CONTACTS AND LOCATIONS:
Locations (1):
- CAIMED, Chía, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: An open-label, balanced, randomized, two treatments, two sequences, four periods, fully replicate, crossover study to evaluate the bioequivalence of Dasatinib 100 mg film-coated tablets of Abbott Laboratories versus Sprycel® (Dasatinib) 100 mg filmcoated — https://www.jscimedcentral.com/Bioavailability/bioavailability-2-1007.pdf